CLINICAL TRIAL: NCT07082881
Title: Impact of Colostrum Oropharyngeal Immunotherapy on Postnatal Growth in Preterm Infants Based on Early Gut Microbiota-Host Interaction Patterns: A Protocol for a Randomized Controlled Trial
Brief Title: Impact of Colostrum Oropharyngeal Immunotherapy on Postnatal Growth in Preterm Infants
Acronym: IOCOIOPGIPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suqian First Hospital (Other)
Responsible Party: Principal Investigator, Na Wang, Principal Investigator, Suqian First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: suqianFH
Record Dates: First submitted 2025-07-05; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Growth Failure; Preterm Birth; Microbiota
MeSH Terms: conditions — Failure to Thrive; Premature Birth | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colostrum Oropharyngeal Immunotherapy (Experimental): The study population will be randomly assigned to either the oropharyngeal colostrum administration group or the normal saline administration group. The intervention will commence within 48-72 h of birth and will be administered continuously for a duration of 5 days, with stool samples collected from the preterm infants before and after the intervention.
  Interventions: Other: Colostrum
- oropharyngeal normal saline administration (Placebo Comparator): The study population will be randomly assigned to either the oropharyngeal colostrum administration group or the normal saline administration group. The normal saline administration will commence within 48-72 h of birth and will be administered continuously for a duration of 5 days, with stool samples collected from the preterm infants before and after thenormal saline administration.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Colostrum — The treatment group will undergo the following treatment protocol within the initial 48-72 h: Investigators will select storage bags with the closest lactation time to the current time while wearing sterile gloves for the entire procedure. Next, using two 1-mL sterile syringes, investigators will draw 0.1 mL of colostrum from each bag and tightly cap the needle hubs to ensure hygiene and safety. Each syringe will be labeled with the hospitalization number, the infant's name, and the date of the mother's colostrum expression. The bags will be then left to sit at room temperature for 5 min to reach an appropriate temperature for oropharyngeal administration of the colostrum. Subsequently, the tip and cap of the first syringe will be removed, and the colostrum will be slowly injected along the right oral mucosa of the participants, lasting at least 20 s. After injection, a sterile cotton swab will be used to gently wipe the right buccal mucosa for at least 10 s.
  Arms: Colostrum Oropharyngeal Immunotherapy
Other: Normal Saline — For the control group, normal saline will be used instead of colostrum. The rest of the procedure will be the same as that for the treatment group.
  Arms: oropharyngeal normal saline administration

SUMMARY:
The goal of this clinical trial is to ascertain whether oropharyngeal administration of colostrum contributes to postnatal growth in very preterm infants (those born before 32 weeks of gestation). The main questions it aims to answer are:

Can Oropharyngeal administration of colostrum effectively lower the incidence rate of extrauterine growth restriction (EUGR) in participants? Does oropharyngeal colostrum intervention bring about changes in the early gut microbiota of participants? Researchers will conduct a comparative analysis between colostrum and a placebo (normal saline) to investigate whether oropharyngeal administration of colostrum has a beneficial effect on the postnatal growth of participants.

Participants will:

Initiation of oropharyngeal colostrum administration will take place within 48 - 72 hours after birth, and the treatment will be administered continuously for a period of 5 days.

Stool samples will be collected from the participants both before and after the intervention.

Participants will be required to maintain a diary to document their basic characteristics and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age <32 weeks and birth weight <1500 g;
2. admitted to the NICU of one of the five hospitals mentioned above within 24 h of birth; and
3. able to initiate the protocol within 72 h of birth and continuously provide adequate colostrum until the end of the protocol.

Exclusion Criteria:

1. Death within 48 h;
2. severe birth asphyxia (defined as umbilical artery/first-hour arterial blood gas pH < 7.0);
3. birth with severe gastrointestinal malformations (e.g., intestinal atresia, tracheoesophageal fistula, malrotation of the intestines, and Hirschsprung's disease);
4. prenatal diagnosis of congenital chromosomal abnormalities or suspected congenital genetic metabolic diseases; and
5. maternal substance abuse or contraindications to breastfeeding (e.g., HIV).

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of extrauterine growth restriction (EUGR) among participants at the time of hospital discharge | The time frame extends from the first day of hospitalization to the day of discharge, covering the entire inpatient stay, with an average duration of 1.5 months.
  EUGR is defined as the situation where the growth measurement (weight, head circumference, or body length) taken at the time of discharge is less than or equal to the 10th percentile of the predicted value based on the Fenton 2013 growth chart.

SECONDARY OUTCOMES:
The inter-group variances in the gut microbiota of participants subsequent to the intervention | The seventh day after birth
  The inter - group variances in alpha diversity of the gut microbiota between the colostrum - treated group and the placebo - treated group after the intervention
Intergroup difference in the time to regain birth weight | Up to 10 days, with an average of 5 days.
  The time to regain birth weight is an easily overlooked variable in the nutritional management of preterm infants. Previous studies have shown a significant linear relationship between the time to regain birth weight and the growth of very preterm infants after birth. Combining the factors of gestational age and birth weight can better reflect the growth of preterm infants after birth and a nutritional evaluation index for a Neonatal Intensive Care Unit.
The incidence rate of bronchopulmonary dysplasia | The time frame extends from the first day of hospitalization to the day of discharge, covering the entire inpatient stay, with an average duration of 1.5 months.
  Bronchopulmonary dysplasia (BPD) is a chronic lung disease that predominantly affects premature infants, especially those with extremely low birth weights or those who have experienced severe respiratory distress syndrome shortly after birth. It represents a significant complication in neonatal intensive care units and has long - term implications for the respiratory health and overall development of affected infants. Here, BPD is defined as the need for oxygen or respiratory support at the corrected gestational age of 36 weeks.

REFERENCES:
- [Derived] Wang N, Hu Y, Qiu W, He M, Zang Q, Wang B, Tang B, Zhang H, Ni P, Zhu S, Zhang J. Impact of colostrum oropharyngeal immunotherapy on postnatal growth in preterm infants based on early gut microbiota-host interaction patterns: protocol for a randomized controlled trial. Int Breastfeed J. 2025 Sep 29;20(1):72. doi: 10.1186/s13006-025-00769-7. PMID 41024070